CLINICAL TRIAL: NCT04822350
Title: AVENANCE - A Non-interventional Study to Provide Real-world Data on the Use of Avelumab as a Maintenance Treatment for Patients With Advanced or Metastatic Urothelial Carcinoma
Brief Title: A NON-INTERVENTIONAL STUDY ON AVELUMAB USE IN PATIENTS WITH ADVANCED OR METASTATIC UROTHELIAL CARCINOMA
Acronym: AVENANCE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: B9991045; NCT04822350 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2021-03-22; First posted 2021-03-30 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Urothelial Carcinoma
Keywords: Avelumab; Non-interventional study; Effectiveness; France; Maintenance; Immunotherapy; Bladder cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — avelumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Locally advanced or metastatic urothelial carcinoma patients treated with avelumab
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — As provided in real world practice

SUMMARY:
A multicenter ambispective (retrospective and prospective) non-interventional study of patients with locally advanced or metastatic urothelial carcinoma (adv/mUC) treated with avelumab in France, not impacting the treatment decision made by the treating physician and the medical management of treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years of age
2. Patient with locally advanced or metastatic urothelial carcinoma (irrespective of tumor histology) whose disease has not progressed (ongoing stable disease, partial response or complete response) following completion of first-line platinum-based chemotherapy and who has been (retrospective), is (retrospective and prospective), will be (prospective) treated with avelumab.

   * For a patient alive at the moment of the inclusion in the study : the patient must be informed of the study, he/she must be given an information letter signed by the investigator and must not be opposed to the collection of his/her data
   * For a patient who died before the inclusion in the study : the patient (during his life time) must not be opposed in writing to the collection of his data.
3. Patient benefiting from a social security scheme according to local regulations

   Exclusion Criteria:
4. For a patient alive at the moment of the inclusion in the study: patient without liberty, under tutelage, or unable to give oral consent.
5. Patient enrolled in a prospective interventional clinical trial assessing an investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced or metastatic Urothelial Carcinoma treated with avelumab as a maintenance treatment
Sampling Method: Probability Sample
Enrollment: 599 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
overall survival | Avelumab initiation up to 4 years
  time between the first injection of avelumab and the date of death from any cause

SECONDARY OUTCOMES:
overall Survival from the start of the chemotherapy used in 1st line | 1st line Chemotherapy start up to 4 years
  time between the first injection of the chemotherapy used in 1st line and the date of death from any cause.
Progression free survival 1 | Avelumab initiation up to 4 years
  time between the first injection of avelumab and the date of progression or death from any cause.
Progression free survival 2 | Avelumab initiation up to 4 years
  time between the first injection of avelumab and the date of progression or death from any cause during the 2nd line of treatment post-avelumab.
overall response rate | Avelumab initiation up to 4 years
  Complete Response or Partial Response as a best response during the avelumab treatment.
duration of response | Beginning of response up to 4 years
  time between the beginning of the response and progression or death from any cause.
duration of treatment | Avelumab initiation up to 4 years
  time between the first and last dose of avelumab.
Patterns of progression under avelumab | Avelumab initiation up to 4 years
  Metastatic sites and type of progression (new lesion(s)/progression of known lesion(s)).
Adverse events (AEs) reporting | Avelumab initiation up to 4 years
  Adverse events (AEs) of any type, grade 3-4 AEs, AEs leading to interruption or discontinuation, AEs leading to death.
Premedications (acetaminophen and antihistamine) | Avelumab initiation up to 4 years
  Proportion of patients who received a premedication at each injection of avelumab. Median number of cycles with premedication.
Patient reported outcome | Initiation of avelumab, 6 weeks, 3 months, and every three months for up to 2 years
  Evolution of PROs NCCN/FACT FBlSI-18 and EQ-5D-5L scores during avelumab treatment.
Overall response rate on subsequent treatments | Discontinuation of avelumab up to 4 years
  Complete Response or Partial Response as a best response during the subsequent treatments
Duration of subsequent treatments | Discontinuation of avelumab up to 4 years
  time between the first and last dose of subsequent treatment
Progression free survival on subsequent treatments | Discontinuation of avelumab up to 4 years
  time between the first dose of subsequent treatment and the date of progression or death from any cause
Overall survival on subsequent treatments | Discontinuation of avelumab up to 4 years
  time between the first dose of subsequent treatment and the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (81):
- France (81):
  - CHU Charles Nicolle, Rouen, Haute-normandie
  - CHU Nantes, Nantes, Pays de la Loire Region
  - Centre Hospitalier du Pays d AIX, Aix-en-Provence
  - CHU Amiens-Picardie, Amiens
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Auxerre, Auxerre
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de la cote Basque, Bayonne
  - Chru Besancon, Besançon
  - Clinique Tivoli-Ducos, Bordeaux
  - CHU de Bordeaux - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier de Boulogne Sur Mer, Boulogne-sur-Mer
  - Centre Hospitalier Regional Universitaire de Brest, Brest
  - Clinique Pasteur - Lanroze, Brest
  - Hopital Louis Pradel, Bron
  - CENTRE HOSPITALIER Dr Jean-Eric TECHER, Calais
  - Medipole de Savoie, Challes-les-Eaux
  - Centre de Lutte Contre Le Cancer - Auvergne Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Universitaire Gabriel Montpied, Clermont-Ferrand
  - Pole Sante Republique, Clermont-Ferrand
  - Polyclinique Saint Come, Compiègne
  - Clinique de Flandre, Coudekerque-Branche
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Centre Leonard de Vinci, Dechy
  - Clinique Clement Drevon, Dijon
  - Centre Hospitalier Intercommunal Louviers, Elbeuf
  - Centre Hospitalier Annecy Genevois, Epargny METZ Tessy
  - Clinique Du Mousseau, Évry
  - Chi Frejus - Saint Raphael, Fréjus
  - Chi Alpes Du Sud, Gap
  - Centre Hospitalier de Grenoble, Greboble
  - Groupe Hospitalier Mutualiste de Grenoble Institut Daniel Hollard, Grenoble
  - Centre Hospitalier Haguenau, Haguenau
  - Polyclinique de Blois, La Chaussée-Saint-Victor
  - La Roche Sur Yon - Centre Hospitalier Departemetal Vendee, La Roche-sur-Yon
  - Groupe Hospitalier La Rochelle - Re - Aunis, La Rochelle
  - Clinique Victor Hugo, Le Mans
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Polyclinique Du Bois, Lille
  - Clinique de la Louvière, Lille
  - Chu Dupuytren Service Oncologie, Limoges
  - Polyclinique de LIMOGE-Clinique François CHENIEUX, Limoges
  - Centre Hospitalier Jura Sud, Lons-le-Saunier
  - Centre Hospitalier Bretagne Sud, Lorient
  - Clinique de la Sauvegarde, Lyon
  - Centre Leon Berard, Lyon
  - Hopital Europeen, Marseille
  - Hopital de La Timone, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Hopital prive Arnault Tzanck, Mougins
  - Centre D'Oncologie de Gentilly, Nancy
  - Hopital prive du Confluent S.A.S, Nantes
  - Clinique Saint Georges, Nice
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancerologie Du Gard, Nîmes
  - ONCOGARD, Nîmes
  - Hopital Prive Sainte Marie, Osny
  - Hopital Saint-Louis, Paris
  - Hopital Pitie Salpetriere, Paris
  - Hopital Cochin/Unité de Cancerologie, Paris
  - Groupe Hospitalier Diaconesse La Croix Saint Simon, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Polyclinique Marzet, Pau
  - Centre Hospitalier de Cornouaille, Quimper
  - Institut Jean Godinot, Reims
  - Centre Hopistalier Roanne, Roanne
  - Ch Roubais, Roubaix
  - Clinique Mathilde, Rouen
  - Centre Hospitalier Prive Saint Gregoire, Saint-Grégoire
  - Hia Begin, Saint-Mandé
  - Clinique mutualiste de l Estuaire, Saint-Nazaire
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Hospitalier de Soissons, Soissons
  - Clinique Sainte Anne, Strasbourg
  - ICANS - Institut de cancerologie Strasbourg Europe, Strasbourg
  - Hopital Foch, Suresnes
  - Hia Sainte Anne, Toulon
  - IUCT - Oncopole, Toulouse
  - Centre Alexis VAUTRIN, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991045